CLINICAL TRIAL: NCT02766660
Title: Optic Disc, Macula, and Retinal Nerve Fiber Layer Measurements Obtained by OCT in Thyroid Associated Ophthalmopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neon Hospital (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-379
Record Dates: First submitted 2016-04-24; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-04

CONDITIONS: Thyroid Associated Ophthalmopathy
Keywords: Thyroid ophthalmopathy; optical coherence tomography
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thyroid ophthalmopathy (Other): Thyroid associated ophthalmopathy patients were measured by optical coherence tomography.
  Interventions: Device: Optical Coherence Tomography
- Control (Other): Control group was consisted by age and sex- macthed healthy people adn they were measured by optical coherence tomography.
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography — All groups were measured by optical coherence tomography.

SUMMARY:
The aim of the study is to compare the measurements of retinal nerve fiber layer (RNFL), macula and optical disc parameters obtained by optical coherence tomography (OCT), and intraocular pressure (IOP) between the patients with thyroid-associated ophthalmopathy (TAO) and healthy controls.

DETAILED DESCRIPTION:
One hundred and thirty two eyes of 66 patients with TAO and 72 eyes of 36 healthy controls were included in the study. Proptosis level was determined by Hertel exophthalmometer. Optic disc, peripapillary retinal nerve fiber layer and macula parameters were measured by OCT. All measurements were compared between the patients and age and sex-matched healthy controls.

ELIGIBILITY:
Inclusion Criteria: Patient group consists the consecutive patients with thyroid associated ophthalmopathy consulted by endocrinology department.

The control group was chosen among healthy volunteers who have

* no eye pathology,
* 20/20 vision (corrected or uncorrected),
* age and sex-matched with the patient group.

Exclusion Criteria:

For both groups, those who had

* significant sight impairment,
* high myopia ( < -5Diopters ),
* high hyperopia ( > +3Diopters ),
* optic disc anomaly,
* vitreoretinal interface disease,
* vascular and degenerative retinal diseases,
* cornea or lens opacity, ocular surgery history,
* glaucoma,
* neurological diseases that can affect the visual field,
* history of trauma, amblyopia,
* diplopia,
* keratitis,
* history of topical or systemic steroid

Ages: 12 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Macular thickness | one year (between Jan 2012 and Jan 2013)
  Macular thickness (micrometer) was measured by optical coherence tomography in patients and controls.
Retinal nerve fiber layer thickness | one year (between Jan 2012 and Jan 2013)
  Retinal nerve fiber layer thickness (micrometer) was measured by optical coherence tomography in patient and control groups.

SECONDARY OUTCOMES:
Optic disc parameters | one year (between Jan 2012 and Jan 2013)
  Optic disc parameters (morphologic structures) were obtained by optical coherence tomography for both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nurşen ARITÜRK, Prof., Principal Investigator — Ondokuz Mayıs University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sayin O, Yeter V, Ariturk N. Optic Disc, Macula, and Retinal Nerve Fiber Layer Measurements Obtained by OCT in Thyroid-Associated Ophthalmopathy. J Ophthalmol. 2016;2016:9452687. doi: 10.1155/2016/9452687. Epub 2016 Jul 17. PMID 27493796